CLINICAL TRIAL: NCT07127367
Title: Treating New Learning and Memory Deficits Following Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-1301-25
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Stoke
Keywords: Memory; Learning; Stroke
MeSH Terms: conditions — Stroke | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KFmSMT (Experimental): Memory training on computer, 2 times per week for 5 weeks
  Interventions: Behavioral: Memory Training
- Memory program (Sham Comparator): Memory training on computer, 2 times per week for 5 weeks
  Interventions: Behavioral: Memory Training

INTERVENTIONS:
Behavioral: Memory Training — Memory retraining exercises will be administered on a laptop computer twice a week for five weeks (10 training sessions).

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a memory enhancement technique in persons following stroke

ELIGIBILITY:
Inclusion Criteria:

* Stroke over 1 year ago
* Memory challenges

Exclusion Criteria:

* Aphasia
* non English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
CVLT-III | baseline, week 7 and 6 months following intervention.
  16 words from 4 semantic categories presented over 5 learning trials. Includes Free and cued immediate and delayed recall and delayed recognition
modified Ecological Memory Simulations (EMS) | Baseline, week 7, and 6 months following intervention
  Everyday memory simulations, recalling a story or directions from a doctor

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berg I, Koning-Haanstra M, Deelman B. Long-term effects of memory rehabilitation: A controlled study. Neuropsychol Rehabil. 1(2):97-111.
- [Background] Gross AL, Rebok GW. Memory training and strategy use in older adults: results from the ACTIVE study. Psychol Aging. 2011 Sep;26(3):503-17. doi: 10.1037/a0022687. PMID 21443356